CLINICAL TRIAL: NCT01751581
Title: The Effect of Sleep Reduction on Daily Energy Expenditure, Thermic Effect of Food, and Substrate Oxidation in Overweight Women
Brief Title: Sleep Restriction and Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SLR-P&F-1
Record Dates: First submitted 2012-06-06; First posted 2012-12-18 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-12

CONDITIONS: Obesity
Keywords: Obesity; Resting Metabolic Rate; Sleep; Eating
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Habitual Sleep (Active Comparator): Women sleep 8 h/night throughout the study phase
  Interventions: Behavioral: Habitual sleep
- Short Sleep (Experimental): Women sleep 4 h/night throughout the study phase
  Interventions: Behavioral: Short Sleep

INTERVENTIONS:
Behavioral: Short Sleep — Participants will be restricted in sleep and only allowed to sleep from 1 am to 5 am.
  Arms: Short Sleep
Behavioral: Habitual sleep — Participants sleep 8 h/night throughout the study phase (from 11 pm to 7 am)
  Arms: Habitual Sleep

SUMMARY:
Each 4-day period will follow the same protocol. Basically, for the entire study, we will prepare all of the subject's food and will require him or her to eat all of the food that we give at the times we tell them to eat. The subject will arrive at the hospital on the evening of day 1, and become inpatients. On day 2, the subject will be permitted to leave the hospital campus under the supervision of the research staff. On day 3, they will be required to stay in a small room called a metabolic chamber for 24 hours. This room measures how many calories you burn in one day. On day 4, we will measure the subject's energy expenditure in response to a breakfast meal. They will be given breakfast and the number of calories that they burn after that meal will be measured over a 6-hour period. Then the subject will be discharged at the end of the test. The 2 study periods will differ only in bedtimes and wakeup times. During one period, the subject will go to bed at 1 am and wake up at 5 am and during the other period they will go to bed at 11 pm and wake up at 7 am.

DETAILED DESCRIPTION:
Sleeping metabolic rate will be measured using a metabolic chamber on the night of day 2. During day 3, 24-hour energy expenditure (including a second night of measurement) will be measured in the metabolic chamber. On this day, the participant will perform 2 bouts of physical activity on a stationary bicycle for 15 minutes each bout. This will give us a measurement of physical activity energy expenditure. On day 4, at 7 am, the participant will exit the metabolic chamber and will enter a different, smaller metabolic chamber for the measurement of energy expenditure in response to a meal. This measurement will start at approximately 8 am with assessment of the resting metabolic rate (45 minutes). The participant will then be given a high-fat meal replacement to consume over 10 minutes. Energy expenditure measurements continue in the metabolic chamber for a 6-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-45 yrs
* Non-pregnant, non-lactating female subjects
* Body mass index (BMI) 25-28 kg/m2
* Weight stable (± 2.5 kg) for at least 3 mo prior to evaluation
* If a woman of child-bearing potential, must be willing to adhere to an acceptable form of contraception
* Non-smoker
* Regularly sleeps 7-8.5 hours/night
* If taking any form of medication, other than those listed in the exclusion criteria, must have been stable and remain on the same medication and medication dose throughout the study

Exclusion Criteria:

* Diabetes, uncontrolled hypertension
* Attempted to lose weight in past 3 months
* Eating disorder
* Stroke, seizure disorder, or other significant neurological disease;
* HIV positive by self-report
* Unstable or uncontrolled medical illness including active malignancies within past 5 yrs
* Untreated or unstable hypothyroidism
* Hyperthyroidism
* A score on the Brief Psychiatric Inventory that exceeds the 90th percentile;
* Subjects with psychoses, bipolar disorder, major depression, severe personality disorders, suicidal
* Alcohol or substance abuse in the past 6 mo
* Pregnant, planning pregnancy in the next 6 mo, or breast-feeding
* Participating in a commercial diet or behavior modification program (e.g., Weight Watchers), or plans to participate
* Shift worker, commercial long-distance driver, heavy equipment operator, history of drowsy driving
* Takes naps regularly
* Has traveled across time zones in the past 4 weeks or plans to during the weeks of the study
* Excessive caffeine intake

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic Rate | 32 hours
  Metabolic rate from 11 pm on day 2 until 7 am on the morning of day 4 will be measured in a metabolic chamber. The metabolic chamber is an air-tight room (22,000 l volume) equipped with a bed, chair, desk, television, VCR, telephone, treadmill, sink and toilet. All meals and snacks will be served at the scheduled time. Subjects will be asked to perform 30 min of light physical activity at 1500 h and 2030 h. Physical activity will consist of 30 min of cycling at 12 mi/h. Bedtimes will be the same as the previous night and actigraph monitoring will be used to confirm compliance with the sleep protocol. Women will exit the chamber at 0700 h the following day.

SECONDARY OUTCOMES:
Post Prandial Energy Expenditure and Thermic Effect of Food | 8 hours on day 4
  Energy expenditure will be measured from 8 am until approximately 2:30 pm on day. Resting metabolic rate over 45 minutes will be measured at 8 am, followed by breakfast and resumption of energy expenditure measurements postprandially.
  Participants will be given 15 min to consume a high-fat breakfast (50% of energy from fat) and post-prandial thermogenesis and substrate oxidation will be measured for the next 6 h.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St. Onge, PhD, Principal Investigator — St. Luke's Roosevelt Hospital/Columbia University
Locations (1):
- St. Luke's Hospital, New York, New York, United States

REFERENCES:
- [Derived] Shechter A, Rising R, Albu JB, St-Onge MP. Experimental sleep curtailment causes wake-dependent increases in 24-h energy expenditure as measured by whole-room indirect calorimetry. Am J Clin Nutr. 2013 Dec;98(6):1433-9. doi: 10.3945/ajcn.113.069427. Epub 2013 Oct 2. PMID 24088722